CLINICAL TRIAL: NCT05114161
Title: Promoting Optimal Treatment for Community-acquired Pneumonia in the Emergency Room (PIONEER): a Prospective, Before-after, Cohort Study
Brief Title: Promoting Optimal Treatment for Community-acquired Pneumonia in the Emergency Room (PIONEER)
Acronym: PIONEER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Jeffrey Pernica, Head, Division of Infectious Disease, Hamilton Health Sciences Corporation
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HAH-20-12
Record Dates: First submitted 2021-10-18; First posted 2021-11-09 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Community-acquired Pneumonia
Keywords: Community-Acquired Pneumonia; Diagnostics; Respiratory Viruses; Mycoplasma
MeSH Terms: conditions — Community-Acquired Pneumonia; Mycoplasma Infections

STUDY DESIGN:
Intervention Model Description: Before-after study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): All participants/caregivers will be asked for consent for point-of-care (POC) blood C-reactive protein (CRP), nasopharyngeal swab for virology/Mycoplasma testing, and urine for pneumococcal antigen (UAg) testing, but, since this testing will not affect care, these are optional (ie. refusal will not preclude enrolment). The RA will phone the caregiver at Day 2-5, Day 14-21, and Day 30 post-enrollment, for outcome ascertainment. Caregivers will be asked to fill out a daily diary (either electronically or on paper) to record the participant's symptoms, clinical progress, and possible drug adverse effects. Caregivers will also be instructed on how to take patient temperature. All participants whose symptoms do not progressively improve will be encouraged to return to the ED to be reassessed, as per standard of care.
- Novel Care Pathway (Experimental): Once a child is diagnosed with non-severe CAP (community-acquired pneumonia) in the ED, specific radiographic findings and point-of-care CRP testing will identify those who require antibiotic treatment immediately. The next day, results of multiplex respiratory pathogen and urine pneumococcal antigen (UAg, optional) testing will be integrated into the care plan, along with additional clinical information about the child gathered remotely, to ensure that only children at appreciable risk for bacterial infection receive antibiotics. Our care pathway uses already-available testing (NPS) in new ways, integrates newer diagnostics (point-of-care CRP, UAg), and includes properly-timed clinical follow up to change how children with non-severe CAP are managed.The research team will follow-up with the participant and caregiver the next day, 2-5 days, 7-21 days and day 30 post-enrolment to ensure clinical stability.
  Interventions: Other: Novel Care Pathway

INTERVENTIONS:
Other: Novel Care Pathway — The novel care pathway will follow a decision tree based on several criteria to stratify patients in an appropriate risk category. Patients with large radiographic lobar consolidation OR POC CRP > 60mg/L will be deemed 'appreciable risk' while patients with CRP < 20mg/L will be deemed 'low risk'. Patients with CRP between 20 - 60mg/L will be evaluated further, as follows: if they have an oxygen saturation of <95%, they will be 'appreciable risk', and if not, there are further decision points: if they are not tachypneic, they will be 'low risk'; if they are tachypneic and less than 1 year of age, they will be 'appreciable risk'; if they are tachypneic, over 1 year of age, but with either complete PCV13 immunization OR detectable wheezing as per the ED clinician, they will be classified as 'low risk'. Appreciable-risk participants will be given a prescription for antibiotics at ED discharge.
  Arms: Novel Care Pathway

SUMMARY:
Pneumonia in children can be caused by different types of germs such as bacteria and viruses. Giving antibiotics to children with bacterial bugs is helpful while giving antibiotics to children with viruses will not help them. Unfortunately, it is difficult for doctors to tell when a child's pneumonia is caused by bacteria or viruses. Most young children are given antibiotics even though it doesn't help them.

Our study wants to test a new way to care for children with pneumonia so that only children who will benefit from antibiotics will receive them. The study will use a combination of the child's symptoms, x-rays results, and lab testing to better determine if a child needs antibiotics. The study team will then review the testing results and follow up with the patient and their family in the following days to ensure that the child is improving. PIONEER will test a novel care pathway for treating non-severe pediatric pneumonia with the goal of decreasing antibiotic prescription while maintaining equal clinical outcomes to standard care.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed primarily with community-acquired pneumonia as per the ED MD and are well enough to be discharged home.
2. They also must have any one of:

   1. tachypnoea;
   2. cough;
   3. increased work of breathing; or
   4. auscultatory findings consistent with pneumonia;

Exclusion Criteria:

Children will be excluded if they have any of the following: cystic fibrosis, anatomic lung disease, bronchiectasis, congenital heart disease (requiring treatment or with exercise restrictions), history of repeated aspiration/velopharyngeal incompetence, malignancy (current or past), immunodeficiency (primary, acquired, or iatrogenic), pneumonia previously (clinically) diagnosed within the past month, or lung abscess diagnosed within the past six months. Children who present with ongoing fever after 4 or more days of beta-lactam therapy active against S. pneumoniae (ie. amoxicillin, amoxicillin-clavulanate, cefprozil, cephalexin, cefadroxil), levofloxacin/moxifloxacin, or doxycycline will not be eligible. Children will not be eligible to participate more than once.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Genders eligible for Study: All
Enrollment: 162 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Treatment with antibiotics for community-acquired pneumonia | Day 0-14
  The proportion of participants who receive antibiotics specifically targeting community-acquired pneumonia will be assessed at follow-up visits (as per participant caregiver report) and compared between phases of the study (control phase and intervention phase)

SECONDARY OUTCOMES:
Clinical cure | Day 14-21
  Cure defined by 1) symptoms improving as per caregiver report, 2) failure to be hospitalized for community-acquired pneumonia, and 3) lack of receipt of additional antimicrobials specifically for the treatment of community-acquired pneumonia
Re-presentation to the ED | Day 0-30
  The number of participants in each phase with unscheduled ED visits before day 30 will be compared.
Treatment with broad-spectrum antibiotic therapy for community-acquired pneumonia | Day 0-30
  The proportion of participants who receive broad-spectrum antibiotics (ie. amoxicillin/clavulanate, cephalosporins, azithromycin, fluoroquinolones) specifically targeting community-acquired pneumonia will be assessed at follow-up visits (as per participant caregiver report) and compared between phases of the study (control phase and intervention phase)
Occurence of drug-related adverse events | Day 0-30
Development of complicated CAP before day 30 | day 0-30
  (i.e. pleural effusion or PICU admission)
Number of days of missed work (caregiver) | Day 14-21
Number of missed days of school/daycare (participant) | Day 14-21
Caregiver satisfaction with the care plan | Day of enrolment, day 2-5, day 14-21 and day 30 follow-up
  This will be measured using a previously validated scale (Likert scale evaluating satisfaction with each of: overall care, doctor's diagnosis, and antibiotic treatment plan)
Failure to achieve clinical cure in those who have CRP<20 mg/L | Day 0-30
Level of serum procalcitonin that effectively rules out the need for antimicrobials | Day 0-30
  (i.e. the level below which 97.5% of participants experience clinical cure without before prescribed antimicrobials)
Treatment with Mycoplasma-active antibiotics for those in whom Mycoplasma is detected | Day 0-14
Unscheduled visits to primary care (eg family MD, nurse practitioner, physician assistant) before day 30 post-enrolment | Day 0-30
Hospitalization for CAP | Day 0-30
Development of complicated CAP (ie pleural effusion or PICU admission) | Day 0-30

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Pernica, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data relating to the primary outcome will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Protocol and SAP will be available after their publication. Outcome data will be made available after study completion and publication.

REFERENCES:
- [Derived] Pernica JM, Kam AJ, Eltorki M, Khan S, Goldfarb DM, Smaill F, Wong J, Ewusie J, Smieja M, Sung M, Mertz D, Thabane L, Loeb M. Novel care pathway to optimise antimicrobial prescribing for uncomplicated community-acquired pneumonia: study protocol for a prospective before-after cohort study in the emergency department of a tertiary care Canadian children's hospital. BMJ Open. 2022 Nov 17;12(11):e062360. doi: 10.1136/bmjopen-2022-062360. PMID 36396301